CLINICAL TRIAL: NCT01177436
Title: PCA-3 Gene Project
Brief Title: Prostate Cancer Antigen 3 (PCA-3) Gene Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-11; 2009-A00567-50
Record Dates: First submitted 2009-10-14; First posted 2010-08-09 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Prostate Cancer; Benign Prostatic Hypertrophy
Keywords: prostate cancer; benign prostatic hypertrophy
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients treated for prostatic pathology (Experimental): Patients treated for prostatic pathology (benign or malign)in the hospital department.
  Interventions: Biological: Taking of urines

INTERVENTIONS:
Biological: Taking of urines — Urine specimens collected by vesical catheterism just before surgery. The dosage of PCA-3 and the analyse of several prostatic markers (genes coding for androgen receptor and steroid alpha-reductase type 1 and 2) will be realized on the samples of urines.

SUMMARY:
Nowadays, prostate cancer screening is largely widespread although it is not recommended yet. This screening includes primarily digital rectal examination and PSA.

Recently, a new specific genetic marker of prostate cancer has been discovered. It is PCA-3 gene.

The main objective is to evaluate prospectively this new marker in patients treated for prostatic pathology (benign or malign) in the department.

DETAILED DESCRIPTION:
Nowadays, prostate cancer screening is largely widespread although it is not recommended yet. This screening includes primarily digital rectal examination and PSA.

The main drawback is the poor PSA specificity. Prostate cancer diagnosis is only histologic diagnosis (mainly by prostate biopsies). However, prostate needle biopsies have a poor rentability and are negative in 60 to 80%. Recently, a new specific genetic marker of prostate cancer has been discovered. It is PCA-3 gene. This gene encodes for RNAm noncoding. So, RNA expression must be assayed by RT-PCR. The main objective is to evaluate prospectively this new marker in patients treated for prostatic pathology (benign or malign) in the department.

PCA-3 assay will be made from urine specimens collected by vesical catheterism just before surgery. Moreover, the investigators will analyse expression of several prostatic markers (genes coding for androgen receptor and steroid alpha-reductase type 1 and 2). The main objective is to improve the prostate cancer diagnosis specificity. Gene expression will be assayed by RT-PCR.

Prostatic cells in urine specimens will be confirmed by assay of PSA gene expression. Normalization of data will be performed using 3 housekeeping genes expression (ß-actin, K-a-1 tubulin and Glyceraldehyde-3-phosphate).

The originality of this clinical study compared to previous reports, consists to two elements. Firstly, all patients included in our study will be operated for a prostate cancer or a BPH. So, the risk to ignore a prostate cancer will be low unlike prostate biopsies made for a prostate cancer screening. Secondly, PCA-3 assay will be coupled with others prostatic specific markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for a prostate cancer or a benign prostatic hypertrophy
* Patients not in state of emergency

Exclusion Criteria:

* Patients with an urinary infection proved bacteriologically
* Patients with a vesical malign disease
* Patients in state of emergency

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the specificity and the sensibility of PCA-3 marker in patients treated for prostatic pathology (benign or malign). | 18 months

SECONDARY OUTCOMES:
To analyse expression of several other prostatic markers (genes coding for androgen receptor and steroid alpha-reductase type 1 and 2)in the aim to improve the prostate cancer diagnosis specificity. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille BASTIDE, Principal Investigator — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France